CLINICAL TRIAL: NCT01194713
Title: Losing Sleep Over Alzheimer's Disease? Effects of Sleep Deprivation on Cerebrospinal Fluid Amyloid-beta Dynamics
Brief Title: Effects of Sleep Deprivation on Cerebrospinal Fluid (CSF) Amyloid-beta (Aβ) Dynamics
Acronym: AWAKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Dr. J. Claassen, Dr. Jurgen Claassen, University Medical Center Nijmegen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AWAKE32920
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Cerebrospinal fluid; Sleep; Abeta
MeSH Terms: conditions — Alzheimer Disease

ARMS (2):
- Sleep deprivation (Active Comparator): 13 subjects will undergo full sleep deprivation
  these subjects are blind to allocation ntil they enter the study center
  Interventions: Behavioral: Sleep deprivation
- Control night (No Intervention): control night of unrestricted sleep in 13 other subjects

INTERVENTIONS:
Behavioral: Sleep deprivation — subjects will undergo one night of full sleep deprivation
  Arms: Sleep deprivation

SUMMARY:
Introduction: Alzheimer's disease (AD) is characterized by neurodegeneration of the brain in the form of neurofibrillary tangles and plaques containing the amyloid-beta protein (Abeta). Recent animal studies have shown that extended wakefulness is associated with increased production of these Abeta proteins and that sleep leads to a marked fall in their production.

Aim: The investigators aim to distinguish a similar effect of sleep disturbance on cerebrospinal fluid (CSF) Abeta levels in humans, which may point out sleep disturbance as an important factor in AD development.

Methods: a study in 26 healthy male volunteers, measuring CSF Abeta levels during a sleep deprivation night and before and after a control night with unrestricted sleep.

Expected results: The investigators expect sleep deprivation to lead to an increase in CSF Abeta levels, as compared to the levels in the control night.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 40-60 years
* Male
* Subject is in good health as established by medical history, physical examination, ECG and laboratory examination
* Laboratory parameters (as described on in section 3.7 screening) should be within the normal ranges as applicable in RUNMC, Nijmegen, or clinically acceptable to the investigator
* Normal sleep behaviour, Pittsburg Sleep Quality index score ≤5
* MMSE 28 or higher
* Medication free

Exclusion Criteria:

* Presence of blood coagulopathy, established by medical history
* Allergy to local anesthetic agents
* Contra-indication for spinal catheter placement: medical history of compression of spinal cord, spinal surgery, skin infection, developmental abnormalities in lower spine
* Subjects who are currently participating in another study or have participated in a clinical study within 30 days, based on their own report about participation history
* Subjects with a history of drug or alcohol abuse
* Subjects who are part of the study staff personnel or family members of the study staff personnel

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Amyloid beta | 6 timepoints during one night of sleep deprivation
  Subjects will undergo one night of sleep deprivation before, during and after which a total of 9 CSF samples (6ml each) will be drawn through a spinal catheter. From these CSF samples Amyloid beta will be analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre Nijmegen, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Ooms S, Overeem S, Besse K, Rikkert MO, Verbeek M, Claassen JA. Effect of 1 night of total sleep deprivation on cerebrospinal fluid beta-amyloid 42 in healthy middle-aged men: a randomized clinical trial. JAMA Neurol. 2014 Aug;71(8):971-7. doi: 10.1001/jamaneurol.2014.1173. PMID 24887018